CLINICAL TRIAL: NCT00609700
Title: Balanced Volume Replacement Therapy With Ringer's Acetate Solution in Burn Injury
Acronym: VoLTRAB
Status: Completed | Type: Observational
Sponsor: Klinikum St. Georg gGmbH (Other)
Responsible Party: Principal Investigator, Armin Sablotzki, MD, prof. Dr. med., Klinikum St. Georg gGmbH
Other Study IDs: EK-BR-35/07-1; EK-BR-35/07-1
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Severe Burn Injury
Keywords: burn injury; volume replacement; Ringer's Lactate solution; Ringer's Acetate solution; volume replacement with crystalloids
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Historical group: patients treated with Ringer's Lactate solution after severe burn injury
- 2: Actual group: patients treated with Ringer's Acetate solution after severe burn injury

SUMMARY:
This observational study compares the influence of Ringer's Lactate solution and Ringer's Acetate solution on organ function scores following severe burn injury.

DETAILED DESCRIPTION:
In the early period following severe burn injury volume replacement with high amounts of crystalloids is necessary. In this study we compare the organ function scores of a historical patient group, treated with Ringer's Lactate solution, with an actual patient population, treated with Ringer's Acetate solution.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years and <80years
* Burned surface area >20% and <70%
* Burn injury < 24 hours
* Agreement to the study procedures

Exclusion Criteria:

* Burned surface area > 70%
* Expected survival time < 24 hours
* Acute or chronic heart failure NYHA III or IV
* Adult respiratory distress syndrome
* Renal failure
* Hepatic failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients within a 24-hours period after severe burn injury
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-12; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change of SOFA-score from day 3 to day 7 after severe burn injury | day3, day7, day28, day60

SECONDARY OUTCOMES:
Changes in electrolyte-balance | day3, day7, day28

CONTACTS AND LOCATIONS:
Overall Officials: Armin R Sablotzki, MD, Principal Investigator — Klinikum St. Georg Leipzig
Locations (1):
- Klinikum St Georg, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Gille J, Klezcewski B, Malcharek M, Raff T, Mogk M, Sablotzki A, Taha H. Safety of resuscitation with Ringer's acetate solution in severe burn (VolTRAB)--an observational trial. Burns. 2014 Aug;40(5):871-80. doi: 10.1016/j.burns.2013.11.021. Epub 2013 Dec 15. PMID 24342121
- See also: Homepage of study site — http://www.sanktgeorg.de